CLINICAL TRIAL: NCT02421081
Title: Effect of Cell Surface Markers Like CD 34 - CD 133 - CD 309 and Lymphoid Cell Distribution on the Wrist Laceration With Radial or Ulnar Arterial Tissue Repair
Brief Title: Effect of Cell Surface Markers and Lymphoid Cell Distribution on the Arterial Tissue Repair (ECLAR)
Acronym: ECLAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ali eray günay, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKCD
Record Dates: First submitted 2015-03-14; First posted 2015-04-20 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Injury of Radial Artery at Wrist and Hand Level; Injury; Ulnar Artery, Hand and Wrist
Keywords: CD34; CD133; CD309; Radial Artery; Ulnar Artery; Lymphoid Cell; blood levels; endothelial progenitor cells; stem cells
MeSH Terms: conditions — Wounds and Injuries | interventions — Anastomosis, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- having arteriel cut (Active Comparator): 30 patients who refer to Erciyes University emergency department because of wrist laceration with radial and/or ulnar artery incision,will be presenting to the study.All patient's flow rate will be evaluated by Doppler ultrasonography before surgery,as well as the healthy side and side of the cuts.Then 5 ml of blood samples will be taken from the systemic circulation,flowcytometric analysis of serum CD34,CD133 and CD309 levels to be measured.Then after patients received surgery,under a microscope using microsurgical techniques and polyamide suture will be held vascular repair.Patients will be assessed by Doppler ultrasonography again 4 weeks after surgery;flow velocity and vessel diameter will be measured at the anastomoses line and patient will be divided to 4 groups. Among these groups serum CD34,CD133,CD309 levels and distribution of lymphoid cells measured by immunohistochemistry; The relationship between the anastomosis opening will be evaluated statistically.
  Interventions: Procedure: vessel microsurgery; Procedure: tendon repair; Procedure: nerve microsurgery
- having tendon cut (Active Comparator): 10 patients having similar age and sex with first group, who refer to Erciyes University emergency department because of wrist laceration without radial or ulnar artery cutting,will be taken to compare with first group.All patient's flow rate will be evaluated by Doppler ultrasonography before surgery,as well as the healthy side and side of the cuts.Then 5 ml of blood samples will be taken from the systemic circulation,flowcytometric analysis of serum CD34,CD133 and CD309 levels to be measured.Then after patients received surgery to repair tendons and/or nerves. Among these groups serum CD34,CD133,CD309 levels and distribution of lymphoid cells measured by immunohistochemistry; and will compare with first group.
  Interventions: Procedure: tendon repair; Procedure: nerve microsurgery
- healthy control (No Intervention): 10 healty having similar age and sex with first group,controls who accept to give blood to determine normal range of serum CD34,CD133 and CD 309 will be taken to compare with first group.All patient's flow rate will be evaluated by Doppler ultrasonography.Then 5 ml of blood samples will be taken from the systemic circulation,flowcytometric analysis of serum CD34,CD133 and CD309 levels to be measured.

INTERVENTIONS:
Procedure: vessel microsurgery — That is a surgery ro repair artery laceration.
  Other Names: anastomosis; artery repair
  Arms: having arteriel cut
Procedure: tendon repair — That is a surgery ro repair tendon cut.
  Arms: having arteriel cut; having tendon cut
Procedure: nerve microsurgery — That is a surgery ro repair median/ ulnar/ radial nerve cut.
  Arms: having arteriel cut; having tendon cut

SUMMARY:
The radial and ulnar artery injuries related with the wrist cut are frequently encountered. There are many factors which are effective on the improvement of these arterial structures was repaired with microsurgical techniques. Recently has begun to focus on neointimal thickening and endothelialization of the role in vascular healing and maturation made on histopathological study. In this study, the radial and ulnar artery laceration repair healing with the microsurgical anastomosis methods on blood CD34, CD133 and CD309 levels of the effect of the distribution of lymphoid cells has been investigated. The investigators think that; thus by demonstrating the positive impact that may arise; autologous endothelial progenitor cells which are obtained in patients; continuation of anastomotic patency undergoing coronary by-pass or the in hemodialysis patients with arteriovenous fistula; also ensuring the re-flow in patients with acute and chronic peripheral arterial occlusion. The investigators believe could be used for the reimplanted tissue in the limb breakage ensuring that survive.

DETAILED DESCRIPTION:
The radial and ulnar arteries cuts that need to be urgently repaired using microsurgical techniques; after treatment failure rate is quite high among the injured. When straight cut repaired with microsurgical instruments under the microscope cut properly; can be obtained close to excellent results. However, there are many factors that impact on the arterial healing. Hypertension, hypotension, age, diabetes mellitus, obesity and female gender has negative effects on the vascular healing. In recent years, positive effects of endothelialization begun to focus on the improvement; and has been shown to endothelialization on the hematopoietic stem cells and endothelial progenitor cells CD34 and CD133 cd309 is effective. CD34 is a type 1 transmembrane protein and is known as the stem cell marker. Proliferative cells and endothelial stem cells play an important role still in the healing process after vascular incisions. These include CD133 (haematopoietic progenitor cells) and CD309 (Vasculoendotelial Growth Factor Receptor 2) is also believed to be effective. These stem cells and proliferating endothelial cells is called collectively endothelial proliferative cells (EPC). Griese et al in a study had been done on rabbits; autologous endothelial cells, obtained from peripheral blood with immunohistochemical methods, were transplanted after carotid artery intimal injury experimentally.The EPC-treated group was observed that increased endothelialization and significantly reduced neointimal hyperplasia, compared to the control group. Kawamoto et al in their study ex vivo; endothelial progenitor cells in the myocardial ischemic group, has been shown to have positive impact on the preservation of left ventricular function. In another clinical study in patients with peripheral arterial disease with ischemic limbs; increase of oxygen carried in the extremities in the study group, decrease in rest pain, increase in walk distance and had an increase in ankle-brachial index.

In the investigators study on the vessel laceration, such as CD 34, CD133 and CD309 endothelial progenitor cells and stem cells in the blood levels will show whether the effects on vascular healing. Results to be obtained; frequently encountered and the relatively high treatment costs and lead to the loss also great labor; myocardial infarction, peripheral arterial disease, ensuring the fistula opening in chronic dialysis patients, provision of limb preservation and vitality of limb replantation will open up new horizons.

ELIGIBILITY:
Inclusion Criteria:

Patients will be chosen

1. Older from 18 year
2. Don't use any medicine

Exclusion Criteria:

1. younger from 18 years
2. Having another illness
3. Using medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
flow velocity of vessel measure with doppler ultrasonography (cm/sn) | flow velocity will measure from lacere arter distal and whole arter; pre surgery, and 4. week after surgery
  the patients will be divided 4 groups with flow velocity
CD 34 - 133 - 309 measurement with immunohistochemical techniques (piece) | 6 hours after trauma
  CD 34 - 133 - 309 levels will be compared between groups
vessel diameter measure with doppler ultrasonography (cm) | vessel diameter will measure from lacere arter distal and whole arter; pre surgery, and 4. week after surgery
  the patients will be divided 4 groups with vessel diameter

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim KARAMAN, docent, Study Director — TC Erciyes University
Locations (1):
- Erciyes University Faculty of Medicine, Melikgazi, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Result] Allon M, Robbin ML. Increasing arteriovenous fistulas in hemodialysis patients: problems and solutions. Kidney Int. 2002 Oct;62(4):1109-24. doi: 10.1111/j.1523-1755.2002.kid551.x. PMID 12234281
- [Result] Glagov S, Zarins C, Giddens DP, Ku DN. Hemodynamics and atherosclerosis. Insights and perspectives gained from studies of human arteries. Arch Pathol Lab Med. 1988 Oct;112(10):1018-31. PMID 3052352
- [Result] Mattsson EJ, Kohler TR, Vergel SM, Clowes AW. Increased blood flow induces regression of intimal hyperplasia. Arterioscler Thromb Vasc Biol. 1997 Oct;17(10):2245-9. doi: 10.1161/01.atv.17.10.2245. PMID 9351396
- [Result] Guzman RJ, Abe K, Zarins CK. Flow-induced arterial enlargement is inhibited by suppression of nitric oxide synthase activity in vivo. Surgery. 1997 Aug;122(2):273-9; discussion 279-80. doi: 10.1016/s0039-6060(97)90018-0. PMID 9288132
- [Result] Dixon BS, Novak L, Fangman J. Hemodialysis vascular access survival: upper-arm native arteriovenous fistula. Am J Kidney Dis. 2002 Jan;39(1):92-101. doi: 10.1053/ajkd.2002.29886. PMID 11774107
- [Result] Szmitko PE, Fedak PW, Weisel RD, Stewart DJ, Kutryk MJ, Verma S. Endothelial progenitor cells: new hope for a broken heart. Circulation. 2003 Jun 24;107(24):3093-100. doi: 10.1161/01.CIR.0000074242.66719.4A. No abstract available. PMID 12821589
- [Result] Werner N, Junk S, Laufs U, Link A, Walenta K, Bohm M, Nickenig G. Intravenous transfusion of endothelial progenitor cells reduces neointima formation after vascular injury. Circ Res. 2003 Jul 25;93(2):e17-24. doi: 10.1161/01.RES.0000083812.30141.74. Epub 2003 Jun 26. PMID 12829619
- [Result] Griese DP, Ehsan A, Melo LG, Kong D, Zhang L, Mann MJ, Pratt RE, Mulligan RC, Dzau VJ. Isolation and transplantation of autologous circulating endothelial cells into denuded vessels and prosthetic grafts: implications for cell-based vascular therapy. Circulation. 2003 Nov 25;108(21):2710-5. doi: 10.1161/01.CIR.0000096490.16596.A6. Epub 2003 Nov 3. PMID 14597586
- [Result] Kawamoto A, Gwon HC, Iwaguro H, Yamaguchi JI, Uchida S, Masuda H, Silver M, Ma H, Kearney M, Isner JM, Asahara T. Therapeutic potential of ex vivo expanded endothelial progenitor cells for myocardial ischemia. Circulation. 2001 Feb 6;103(5):634-7. doi: 10.1161/01.cir.103.5.634. PMID 11156872
- [Result] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713